CLINICAL TRIAL: NCT01142544
Title: Acute Lung Injury in Children: Epidemiology and Natural History: The Pediatric ALIEN Study
Brief Title: Incidence of Acute Lung Injury in Children
Acronym: PED-ALIEN
Status: Completed | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: Asociación Científica Pulmón y Ventilación Mecánica (Other)
Responsible Party: Principal Investigator, Jesus Villar, Director of Research, Dr. Negrin University Hospital
Other Study IDs: 2010-0915-PED-ALI
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Acute Lung Injury; Children
Keywords: acute lung injury; incidence; lung damage; PaO2/FiO2 ratio
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pediatric ALIEN: All children from 1 month to 18 years old meeting the American-European Consensus Conference definition of acute lung injury
  Interventions: Other: Evaluation oxygenation under standard ventilator settings

INTERVENTIONS:
Other: Evaluation oxygenation under standard ventilator settings — Measure of PaO2 under standard FiO2-PEEP

SUMMARY:
Acute lung injury in children is a syndrome of rapid onset of acute respiratory failure and require admission into intensive care units (ICU) for advanced life support. There are almost no information on epidemiology of acute lung injury. Published studies do not have information for an entire year and none of them have evaluated the degree of oxygenation failure under standard ventilator settings. The investigators will perform a 1-year prospective audit of all patients admitted with acute lung injury in a network of pediatric ICUs in Spain.

DETAILED DESCRIPTION:
We will evaluate oxygenation under standard ventilator settings (FiO2 0.5 and 1 on PEEP 5 or 10 cmH2O) in pediatric acute respiratory distress syndrome.

Outcome measures will include: overall ICU mortality, number of patients meeting ARDS criteria at 24 hours, and stratification of patients depending on PaO2/FiO2 ratio at 24 h of meeting acute respiratory distress syndrome criteria.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset of respiratory failure
* Age 1 month to 18 years old
* Bilateral pulmonary infiltrates on Chest X-ray
* Absence of left ventricular failure, PaO2/FiO2>300 mmHg

Exclusion Criteria:

* None

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children from 1 month to 18 years old, admmitted into ICU, and meeting the American-European Consensus Conference definition for acute lung injury (ALI).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of cases of acute lung injury per 100,000 population | 1 year

SECONDARY OUTCOMES:
Assessment of degree of lung severity at onset and at 24 h of the onset of acute lung injury | 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar, MD, PhD, Principal Investigator — Hospital Dr. Negrin, Las Palmas de Gran Canaria, Spain; Robert M Kacmarek, RRT, PhD, Principal Investigator — Massachusetts general Hospital, Boston USA; Yolanda López, MD, PhD, Principal Investigator — Hospital de Cruces, Barakaldo, Vizcaya, Spain; Amelia Martínez, MD, PhD, Principal Investigator — Hospital Infantil del Niño Jesús, Madrid, Spain
Locations (1):
- Jesús Villar, Las Palmas de Gran Canaria, Las Palmas, Spain

REFERENCES:
- [Derived] Lopez-Fernandez Y, Azagra AM, de la Oliva P, Modesto V, Sanchez JI, Parrilla J, Arroyo MJ, Reyes SB, Pons-Odena M, Lopez-Herce J, Fernandez RL, Kacmarek RM, Villar J; Pediatric Acute Lung Injury Epidemiology and Natural History (PED-ALIEN) Network. Pediatric Acute Lung Injury Epidemiology and Natural History study: Incidence and outcome of the acute respiratory distress syndrome in children. Crit Care Med. 2012 Dec;40(12):3238-45. doi: 10.1097/CCM.0b013e318260caa3. PMID 22990455